CLINICAL TRIAL: NCT03379077
Title: Implementing Learning Through Play (LTP) Plus Group Cognitive Behaviour Therapy (CBT) for Mothers of Young Children (0-3 Years) in Gadap Town (Roshni-2).
Brief Title: Learning Through Play (LTP) Plus Group Cognitive Behaviour Therapy for Mothers of Young Children (ROSHNI-2)
Acronym: ROSHNI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Health and Nutrition Development Society (Unknown); Hincks Dellcrest Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PILL-ROSHNI2
Record Dates: First submitted 2017-12-08; First posted 2017-12-20 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Mothers
Keywords: Mothers; young children; Implementation; Learning through play Plus; Cognitive Behavior Therapy
MeSH Terms: interventions — Long-Term Potentiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: researchers doing outcome assessment will be kept blind on both implementation groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP Plus Supported Implementation (Experimental): LTP Plus Supported Implementation group participants will receive intervention by trained LHWs of HANDS, co-facilitated and supervised by senior trained PILL researchers, expert in delivering LTP plus intervention
  Interventions: Behavioral: LTP Plus
- LTP Plus (Active Comparator): Participants in LTP Plus arm will receive LTP plus intervention by trained LHWs of Health and Nutrition Development Society (HANDS).
  Interventions: Behavioral: LTP Plus

INTERVENTIONS:
Behavioral: LTP Plus — LTP Plus is comprised of two components; Learning through play (LTP) and Cognitive Behavior Therapy (CBT). The LTP Plus is a low-literacy, sustainable program intended to provide parents with information on the healthy growth and development of their young children. The LTP research-based activities enhance children's development while simultaneously promoting attachment security through building parents' ability to read and be sensitive to their children's cues and through active involvement in their children's development. Plus the Thinking Healthy Program (THP) which adopts 'here and now' problem-solving approach. THP uses cognitive behavior therapy (CBT) techniques of active listening, changing negative thinking, and collaboration with the family.
  Other Names: Psycho-social Intervention

SUMMARY:
The study has both quantitative and qualitative components.

The objective of the quantitative study is to:

Determine if supported implementation of the LTP plus programme improves infant development compared to standard implementation of the LTP plus programme.

The objective of the qualitative study is:

Process evaluation and finding out about implementation challenges (from the perspective of the mothers and the people delivering both the LTP plus and the supported implementation intervention).

DETAILED DESCRIPTION:
In Pakistan, the Learning through Play parenting program was tested initially through a cluster randomized study in a rural area of Pakistan. The results of this recently completed cluster RCT funded by the Grand Challenges Canada (GCC) showed that LTP Plus works and benefits both the mother and the child. More specifically, the results indicate a significant reduction in maternal depression.

Purpose of this cluster RCT is to determine if supported implementation of the LTP plus programme improves infant development compared to standard implementation of the LTP plus programme. This is an implementation trial comparing two ways of introducing LTP plus. A Cluster RCT of culturally adapted intervention LTP Plus will be conducted in the villages of Gadap town, Karachi, Pakistan. Total 60 villages will be randomized in two groups LTP plus and LTP plus supported implementation. Each cluster will be made of up to 15 mothers. Participants will be screened using eligibility checklist. Assessments will be done at baseline and after completion of intervention (3-month). All follow ups will be done by independent RAs, not involved in delivering intervention sessions.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if they are:

18 to 44 years old mothers with children aged between 0-33 months, resident in the trial site catchments area, who are able to complete assessments

Exclusion Criteria:

Participants will be excluded from the study if they have:

A medical disorder that would prevent participation in clinical trial. Temporary resident unlikely to be available for follow up. Active suicidal ideation or any other severe or physical mental disorder.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1006 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Infant development: Ages and Stages Questionnaire (Squires, Bricker, & Twombly, 2009) | Change from baseline at 3rd Month
  This scale will be used to measure child development. Parents will report on their child's communication,gross motor, fine motor, problem solving and personal-social development.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ) | Baseline and 3rd Month
  The Patient health Questionnaire (PHQ) is a simple 10 item self-report questionnaire will also be administered by a trained research worker. A score of 10 or more is taken as cut -off for depressive disorder, however all mothers meeting eligibility criteria will be included, despite their scores on PHQ-9.
Generalized Anxiety Disorder (GAD) 7 | Baseline and 3rd Month
  The GAD-7 is a 7 item scale will be used to screen for and measure severity of Generalized Anxiety Disorder
Knowledge of Expectation and Child Development | Baseline and 3rd Month
  A 25-item questionnaire will be used to assess maternal knowledge and expectations for child development in the first three years
Parenting Stress Index - Short Form | Baseline and 3rd Month
  Parents rate 36 items on a five-point scale (1-5) on three scales: (1) Parenting Distress, (2) Difficult Child Characteristics, and (3) Dysfunctional Parent-Child Interaction.
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline and 3rd Month
  This brief scale will be used to measure social support
Euro-Qol-5 Dimensions (EQ-5D) | Baseline and 3rd Month
  Health-related quality of life will be measured using the EQ-5D
Client Service Receipt Inventory | Baseline and 3rd month
  We will collect information about the use of other health services (including the informal sector faith healers/Imams) using CSRI.
CSQ Client Satisfaction Questionnaire | 3rd Month
  The participants will rate their satisfaction with treatment after completion of intervention using the CSQ.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, (MRC Psych, FRC Psych, MD), Principal Investigator — Pakistan Institute of Living & Learning; Nusrat Husain, (MD), Principal Investigator — University of Manchester; Tayyeba Kiran, MS, Principal Investigator — Pakistan Institute of Living & Learning
Locations (1):
- Gadap, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No